CLINICAL TRIAL: NCT00112385
Title: A Pilot Study of Etanercept in Dermatomyositis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Amgen (Industry)
Responsible Party: Anthony A. Amato, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01NS049639-01A2 (NIH); 1R01NS049639-01A2 (NIH); NCT00282880 (obsolete NCT alias)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2011-06-21 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-05

CONDITIONS: Dermatomyositis
Keywords: dermatomyositis; etanercept; tumor necrosis factor alpha
MeSH Terms: conditions — Dermatomyositis | interventions — Etanercept; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etanercept (Active Comparator): Subjects randomized to Etanercept will be provided with syringes contain 50 mg and will be injected subcutaneously once a week for 52 weeks.
  Interventions: Drug: Etanercept
- Placebo (Placebo Comparator): Subjects will be given syringes containing placebo. Injections will be given subcutaneously, one time per week for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etanercept — Etanercept 50 mg will be injected subcutaneously once per week for 52 weeks
  Arms: Etanercept
Drug: Placebo — Placebo, contained in 50mg syringes, will be injected subcutaneously once per week for 52 weeks.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The purpose of the study is to obtain preliminary data regarding the safety and tolerability of etanercept in DM. In addition, we will use the study to assess the variability, reliability, and responsiveness of the core set of outcome measures recommended by IMACS. The study will be performed under the aegis of the Muscle Study Group (MSG), consisting of experienced investigators with an avid interest in myopathies. The ultimate goal of this pilot study will be to obtain necessary, prerequisite information important in designing future therapeutic trials of etanercept and other agents in patients with DM. The specific aims of the study are:

Aim 1: To preliminarily assess the safety and tolerability of etanercept in patients with DM.

Aim 2: To assess the safety and tolerability of prednisone in the dosing schedule we propose to use.

Aim 3: To evaluate outcome measures recommended by IMACS and assess their variability, reliability, and responsiveness in order to facilitate the design of future therapeutic trials in the inflammatory myopathies.

DETAILED DESCRIPTION:
Dermatomyositis (DM) is one of the major subtypes of idiopathic inflammatory myopathy. Prednisone is the initial treatment of choice in most patients with DM. However, because of the high rate of patients with disabling weakness despite treatment with prednisone, the long-term side effects of prednisone, and the many side effects associated with other second-line immunosuppressive agents (e.g., methotrexate, azathioprine), better treatment options are needed. There is evidence that tumor necrosis factor-a (TNF-a) plays a role in the pathogenesis of DM. Thus, etanercept, which blocks TNF-a, is a logical drug to assess in DM. Etanercept has been associated with a number of side effects including an increased risk of infection, inducing other autoimmune diseases, and perhaps cancer. These risks may be further enhanced in DM in which the frequency of other autoimmune disorders (e.g., connective tissue disease) and malignancy are already increased.

The goal of this pilot study will be to assess the safety and tolerability of etanercept in DM.We will perform a double-blind, placebo-controlled pilot study of etanercept in 40 patients with DM randomized in a 3:1 ratio to receive etanercept or placebo. All newly diagnosed and untreated patients will be started on a standard dose of prednisone and tapering schedule. Refractory patients who have been or are currently being treated with prednisone, IVIG, or methotrexate can also participate. Subjects will be followed for 1 year and we will assess various outcome variables recommended by the The International Myositis Assessment Clinical Study Group (IMACS). The primary aim of the study is to preliminarily assess the safety and tolerability of etanercept in patients with DM. We hypothesize that etanercept will be safe and well tolerated in this population. The second aim is to assess the safety and tolerability of prednisone in the dosing schedule we propose to use. We hypothesize that most patients will be able to tolerate the reduction of the prednisone dosage but most will not be able to be completely weaned off the medication. We believe we will find a relationship between prednisone dosage and its related side effects. The third aim of the study is to assess the variability, reliability, and responsiveness of the outcome measures recommended by IMACS using this pilot study of etanercept as the vehicle. The information gained from this study is necessary in order to design larger therapeutic trials of etanercept and other drugs in dermatomyositis.

ELIGIBILITY:
Inclusion Criteria:

Study subjects must meet the following criteria:

1. Meet the diagnostic criteria for DM (a-c; a,b,d; or a,c,d)

   1. Subjects must have symmetric proximal greater than distal weakness
   2. Characteristic DM rash consisting of any or all of the following: heliotrope, shawl sign, V-sign, Gottron's sign, Gottron's papules, periungual telangiectasias
   3. Laboratory evidence of myopathy with at least one of the following: an elevated serum CK or aldolase level, myositis-specific antibody, electromyography (EMG) demonstrating myopathic features (e.g., muscle membrane instability, myopathic units, or early recruitment), or an abnormal skeletal muscle MRI showing diffuse or patchy edema within the muscles.
   4. A muscle biopsy will be optional if the patient fulfills criteria a-c. The subject must demonstrate symmetric proximal weakness (criteria a) for entry into the study. If the subject does not have a definite rash (criteria b) or laboratory evidence of a myopathy (criteria c), a muscle biopsy will be required. The muscle biopsy must demonstrate one of the following: perifascicular atrophy, expression of MHC 1 on perifascicular muscle fibers, MAC deposition on small blood vessels, tubuloreticular inclusions in endothelial cells on EM, or MXA expression on muscle fibers of blood vessels
2. Newly diagnosed subjects should be able to walk independently 30 feet (cane, walkers, orthoses allowed). However, subjects with refractory dermatomyositis may be non-ambulatory.
3. Age > 18 years
4. Patients must not use topical skin ointments for treatment of the dermatological manifestations as it will interfere with skin assessment.
5. Men and women of childbearing age must be willing to use a method of birth control.
6. Able to give informed consent
7. Subject or designee must have the ability to self-inject investigational product or have a care giver at home who can administer subcutaneous injections

Exclusion Criteria

The presence of any of the following excludes subject participation in the study:

1. Presence of any one of the following medical conditions: active infection, uncontrolled diabetes mellitus, MI, CVA or TIA within 3 months of screening visit, symptomatic cardiomyopathy (congestive heart failure), symptomatic coronary artery disease, uncontrolled hypertension (sitting systolic BP <80 mm Hg or > 160 or diastolic BP > 100 mm Hg), oxygen-dependent severe pulmonary disease, systemic lupus erythematosus (SLE), cancer (other than basal cell skin cancer) less than 5 years previously, HIV or other immunosuppressing disease, positive PPD test or any history of mycobacterial disease, chronic hepatitis B or hepatitis C, history of multiple sclerosis, transverse myelitis, optic neuritis, chronic inflammatory demyelinating neuropathy, epilepsy, or other chronic serious medical illnesses
2. Presence of any of the following on routine blood screening: WBC<3000, Platelets < 100,000, hematocrit < 30%, BUN > 30 mg %, symptomatic liver disease with serum albumin < 3 G/DL, PT or PTT > upper range of control values
3. Forced Vital Capacity < 50% of predicted
4. History of non-compliance with other therapies
5. Any prior or concurrent cyclophosphamide, or current use of any immunosuppressive agent besides methotrexate (e.g., azathioprine, mycophenolate, or cyclosporine)
6. Coexistence of other neuromuscular disease that may complicate interpretation of the results of the study
7. Drug or alcohol abuse within last 3 months
8. Pregnancy or breast feeding
9. Juvenile DM
10. Subjects who have known hypersensitivity to Enbrel or any of its components or who is known to have antibodies to etanercept
11. Use of a live vaccine 90 days prior to, or during this study.
12. Subject is currently enrolled in another investigational device or drug trial(s), or subject has received other investigational agent(s) within 28 days of baseline visit.
13. Concurrent sulfasalazine therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony A Amato, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Muscle Study Group. A randomized, pilot trial of etanercept in dermatomyositis. Ann Neurol. 2011 Sep;70(3):427-36. doi: 10.1002/ana.22477. Epub 2011 Jun 17. PMID 21688301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 153 patients were screened and we enrolled and randomized 16 subjects (F 10, M 6) from until February 2006 to May 2009. Of these, 5 were new DM patients and 11 were refractory dermatomyositis patients.
  Etanercept: 11 subjects (New 3, Refractory 8) Placebo: 5 subjects (New 2, Refractory 3)
Pre-assignment Details: Most patient were initially ineligible because they were not new dermatomyositis patients.
  Due to slow recruitment, we modified the protocol. We allowed enrollment of refractory dermatomyositis patients receiving prednisone for greater than 2 months. These subjects could also receive second line agents, as long as they were on a stable dose.
Groups:
- Etanercept: Subjects randomized to Etanercept will be provided with syringes contain 50 mg and will be injected SQ once a week for 52 wks
- Placebo: Subjects will be given syringes containing placebo
Period: Overall Study
Arm/Group | Etanercept | Placebo
Started | 11 | 5
Completed | 10 | 4
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept | Placebo | Total
Number analyzed (Participants) | 11 | 5 | 16
Age Categorical [Number; unit: participants]
  < 18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 5 | 16
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.36 (14.8) | 44.2 (11.9) | 43.6 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 1 | 1
  United States | 11 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of at Least One Adverse Event
Description: Adverse events (AEs) were assessed using the Common Terminology Criteria for Adverse Events version 3.0 (CTCAE). The grade of "mild", "moderate" or "severe" matches with the descriptions from the CTCAE dictionary.
  In general, a "Mild" AE is asymptomatic; clinical or diagnostic observations only; intervention not indicated.
  A "Moderate" AE is minimal, local or noninvasive intervention indicated; limiting activities of daily living.
  A "Severe" AE is medically significant but not immediately life-threatening; hospitalization or prolonged hospitalization indicated; disabling;
Time Frame: at each visit during the 12 month study
Population: Intention- to -Treat (ITT)
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants
  Mild AE | 1 | 1
  Moderate AE | 5 | 1
  Severe AE | 5 | 3

2. Other Pre Specified Outcome: The Number of Participants Who Were Classified as Treatment Failures
Description: Treatment failures were determined based on criteria from the study protocol using objective and subjective ratings from the study physician. If the study physician felt that the rate of prednisone taper needed to be reduced, the prednisone dose needed to be increased or restarted, or a second-line agent added, the patient will be considered to be a treatment failure.
Time Frame: At any point during the 52 week study
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 6 | 5

3. Secondary Outcome: Average Prednisone Dosage After Week 24
Description: We calculated the average dosage of prednisone from the week 24 visit until the end of the study (week 52).
Time Frame: from week 24 to 52
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
mg | 1.2 [0 to 14.31] | 29.2 [12.65 to 31.39]

4. Other Pre Specified Outcome: Change in the Average Manual Muscle Testing (MMT) Score From Baseline to Week 52
Description: The Manual Muscle Test (MMT) assesses 26 muscle groups. The muscle strength of each muscle group is graded. The score for each muscle group ranges from 0 (No contraction palpable) to 5 (normal strength). The minimum total MMT score is a 0. The maximum total MMT score is a 130.
  The average change in the average Manual Muscle Testing (MMT)from Baseline to Week 52 was calculated. The average score is composed of 26 muscle groups that were tested. The average change was determined by subtracting the Baseline test results from the Week 52 results (Week 52- Baseline).
Time Frame: At Baseline (Week 0) and Week 52
Population: Data for all subjects enrolled in the trial are not available for this assessment. One subject in the placebo group left the study before the Week 52 visit. One subject in the etanercept group was lost to follow-up before the Week 52 visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 10 | 4
Units on a scale | 0.24 (0.29) | 0.30 (0.21)

5. Primary Outcome: Tolerability
Description: The reported tolerability measure was defined as the number of participants that completed the entire 52 week study on their originally assigned treatment.
Time Frame: At any point between Baseline (week 0) and the end of the study (Week 52)
Measure: Number; unit: Participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
Participants | 10 | 4

6. Other Pre Specified Outcome: Average Change in Time to Rise From a Chair From Baseline to Week 52
Description: The Average change in time to rise from a chair comparing Baseline performance to Week 52.The average change was determined by subtracting the Baseline test results from the Week 52 results (Week 52- Baseline).
  This measure was also collected as part of the study protocol at Week 4, 8, 12, 16, 20, 24, 32 and 40.
Time Frame: At Baseline (Week0) and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 10 | 4
Seconds | -.05 (2.64) | -1.22 (1.98)

7. Other Pre Specified Outcome: Average Change in Time (Seconds) to Walk 30 Feet Comparing Performance at Baseline to Week 52
Description: Average change in time to walk 30 feet comparing Baseline performance to Week 52.The average change was determined by subtracting the Baseline test results from the Week 52 results (Week 52- Baseline).
  This measure was also collected as part of the study protocol at Week 4, 8, 12, 16, 20, 24, 32 and 40.
Time Frame: At Baseline (Week0) and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 10 | 4
Seconds | -2.26 (4.81) | -0.55 (1.44)

8. Other Pre Specified Outcome: Average Change in Z-score for Dual-emission X-ray Absorptiometry (DEXA) of the Femur From the Screening Visit to Week 52
Description: The average change in z-score for Dual-emission X-ray absorptiometry (DEXA) of the femur from the Screening visit to the Week 52 visit was calculated. The average change was determined by subtracting the Screening Visit test results from the Week 52 results (Week 52- Screening visit).
  The Screening visit was conducted within 8 weeks of the Baseline visit.
Time Frame: Screening and Week 52
Population: Data for all subjects enrolled in the trial are not available for this assessment. One subject in the placebo group left the study before the Week 52 visit. One subject in the etanercept group was lost to follow-up before the Week 52 visit.
  In addition, data may be missing due to the subject's refusal to complete an assessment or examiner error.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 7 | 4
Z-score | 0.17 (0.48) | -0.57 (0.90)

9. Other Pre Specified Outcome: Average Change in Z-score for Dual-emission X-ray Absorptiometry (DEXA) of the Lumbar Spine From the Screening Visit to Week 52
Description: The average change in z-score for Dual-emission X-ray absorptiometry (DEXA) of the lumbar spine was calculated comparing the results from the Screening visit to Week 52. The average change was determined by subtracting the Screening Visit (Week <8)test results from the Week 52 results (Week 52- screening Visit). The Screening visit occurred within 8 weeks of the Baseline visit.
Time Frame: Screening visit and Week 52.
Population: Data for all subjects enrolled in the trial are not available for this assessment. One subject left the study early and one subject was lost to follow-up before the Week 52 visit. In addition, data may be missing due to the subject's refusal to complete an assessment or examiner error.
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 7 | 4
Z-Score | -0.10 (0.57) | 0.07 (1.01)

10. Other Pre Specified Outcome: Average Change in Physician Global Activity Assessment From Baseline to Week 52
Description: Average change in Physician Global Activity Assessment score from Baseline to Week 52. The assessment used a Visual Analog Scale to rate the subject's global (overall) disease activity. A score of 0 cm indicated no evidence of disease activity. A score of 10.0 cm indicated extremely active disease. The average change was determined by subtracting the Baseline test results from the Week 52 results (Week 52- Baseline).
  This measure was also collected as part of the study protocol at Week 4, 8, 12, 16, 20, 24, 32 and 40.
Time Frame: At Baseline (Week0) and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 10 | 4
cm | -2.36 (2.12) | -1.32 (2.41)

11. Other Pre Specified Outcome: Average Change in Patient Global Activity Assessment Score From Baseline to Week 52
Description: Average change in Patient Global Activity Assessment score from Baseline to Week 52. The assessment used a Visual Analog Scale to rate the subject's perceived global (overall) disease activity. A score of 0 cm indicated no evidence of disease activity. A score of 10.0 cm indicated extremely active disease.
  This measure was also collected as part of the study protocol at Week 12, 24, 32 and 40.
Time Frame: At Baseline (Week0) and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 10 | 4
cm | -2.34 (2.97) | -0.38 (2.76)

12. Other Pre Specified Outcome: Average Change in Cutaneous Disease Activity and Severity Index (CDASI) Score From Week 52 to Baseline
Description: Average change in Cutaneous Disease Activity and Severity Index (CDASI) score from Baseline to Week 52. The assessment graded the severity of the subject's rash. The rash was rated using a a 4-point scale with a score of 0 indicating no rash. The score was added together using all 13 anatomical locations included on the assessment. The average change was determined by subtracting the Baseline test results from the Week 52 results (Week 52- Baseline).
  This measure was also collected as part of the study protocol at Week 4, 8, 12, 16, 20, 24, 32 and 40.
Time Frame: At Baseline (Week0) and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 10 | 4
Units on a scale | -3.05 (4.84) | -0.25 (4.84)

13. Other Pre Specified Outcome: Change in Pruritis Rating From Baseline to Week 52
Description: This is the average change in pruritis score from Baseline to Week 52. The assessment used a Visual Analog Scale to rate the subject's perceived level of pruritis (itchiness). A score of 0 cm indicated "Not itchy at all". A score of 10.0 cm indicated "Extremely itchy".
  This assessment was also completed at Week 4, 8, 12, 16, 20, 24, 32 and 40.
Time Frame: At Baseline (Week0), and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 10 | 4
cm | 0.33 (2.63) | -1.64 (1.69)

14. Other Pre Specified Outcome: Change in Health Assessment Questionnaire (HAQ) Score From Baseline to Week 52
Description: The Health Assessment Questionnaire (HAQ)was completed by subjects to assess the affects of their illness on the ability to function in daily life. The HAQ consists of 8 sections. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do).The 8 scores of the 8 sections are summed and divided by 8. A higher score indicates more impairment.
  The average change was determined by subtracting the Baseline test results from the Week 52 results (Week 52- Baseline).
  This measure was also collected as part of the study protocol at Week 12, 24, 32 and 40.
Time Frame: At Baseline (Week0) and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 10 | 4
Units on a scale | -0.33 (0.45) | -0.34 (0.68)

15. Other Pre Specified Outcome: Forced Vital Capacity (FVC) Average Change in Percent Predicted From Screening to Week 52.
Description: The average change in percent predicted Forced Vital Capacity (FVC) from the Screening Visit to Week 52 was calculated. The average change was determined by subtracting the Screening Visit results from the Week 52 results (Week 52- Screening Visit). The Screening visit occurred within 8 weeks prior to the Baseline visit.
  This assessment was also completed at the Week 24 visit.
Time Frame: Screening Visit and Week 52.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent predicted
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 9 | 4
Percent predicted | -2.56 (8.93) | -1.00 (16.47)

16. Other Pre Specified Outcome: Average Change in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) From the Screening Visit to Week 52
Description: The average change in percent predicted Forced Expiratory Volume in 1 second (FEV1) from Screening to Week 52 was calculated. The average change was determined by subtracting the Screening Visit results from the Week 52 results (Week 52- Screening visit). The Screening visit occurred within 8 weeks prior to the Baseline visit.
  This assessment was also completed during the Week 24 visit.
Time Frame: Screening Visit and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent predicted
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 9 | 4
Percent predicted | -0.67 (11.92) | -4.25 (14.80)

17. Other Pre Specified Outcome: Average Change in Percent Predicted Diffusion Capacity (DLCO)From the Screening Visit to Week 52
Description: Average change in percent predicted Diffusion Capacity (DLCO)from the Screening Visit to Week 52 was calculate. The average change was determined by subtracting the Screening test results from the Week 52 results (Week 52- Screening Visit). The Screening visit occurred within 8 weeks prior to the Baseline visit.
  This assessment was also completed during the Week 24 visit.
Time Frame: Screening visit and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent predicted
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 8 | 3
Percent predicted | -4.50 (14.34) | -14.67 (8.33)

18. Primary Outcome: Average Change in Oral Temperature From Baseline to Week 52
Description: The subject's oral temperature was measured in degrees Celsius. The average change was determined by subtracting the Baseline Visit (Week 0) results from the Week 52 results (Week 52- Baseline (Week 0)).
  This measure was also collected as part of the study protocol at the Screening visit and Week 4,8,12,16,20,24,32 and 40.
Time Frame: At Baseline (Week 0) and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 9 | 4
degrees Celsius | 0.16 (0.64) | 0.20 (0.22)

19. Primary Outcome: Average Change in Respiration Rate From Baseline to Week 52
Description: The subject's respiration rate was measured as number of breaths per minute. The average change was determined by subtracting the Baseline Visit (Week 0) results from the Week 52 results (Week 52- Baseline (Week 0)).
  This measure was also collected as part of the study protocol at the Screening visit and Week 4,8,12,16,20,24,32 and 40.
Time Frame: At Baseline (Week0) and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 9 | 4
breaths per minute | -2.44 (3.17) | -2.00 (4.32)

20. Primary Outcome: Average Change in Systolic Blood Pressure From Baseline to Week 52
Description: The subject's systolic blood pressure was measured in millimeters of mercury (mmHg). The average value was calculated per treatment group for the Baseline and Week 52 visit based on treatment group. The average change was determined by subtracting the average value Baseline Visit (Week 0) results from the Week 52 results (Week 52- Baseline (Week 0)).
  This measure was also collected as part of the study protocol at the Screening visit and Week 4,8,12,16,20,24,32 and 40.
Time Frame: At Baseline (Week0) and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 10 | 4
mmHg | -13.3 (16.3) | -3.0 (14.72)

21. Primary Outcome: Average Change in Diastolic Blood Pressure Comparing Baseline to Week 52.
Description: The subject's diastolic blood pressure was measured in millimeters of mercury (mm Hg). The average value was calculated for the Baseline and Week 52 visit based on treatment group. The average change was determined by subtracting the average value Baseline Visit (Week 0) results from the Week 52 results (Week 52- Baseline (Week 0)).
  This measure was also collected as part of the study protocol at the Screening visit and Week 4,8,12,16,20,24,32 and 40.
Time Frame: At Baseline (Week0) and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 10 | 4
mmHg | -6.10 (9.52) | 1.00 (7.39)

22. Primary Outcome: Average Change in Pulse Comparing Baseline to Week 52
Description: The subject's pulse was measured in beats per minute (BPM). The average value was calculated per treatment group for the Baseline and Week 52 visit. The average change was determined by subtracting the average value Baseline Visit (Week 0) results from the Week 52 results (Week 52- Baseline (Week 0)).
  This measure was also collected as part of the study protocol at the Screening visit and Week 4, 8, 12, 16, 20, 24, 32 and 40.
Time Frame: At Baseline (Week0) and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 10 | 4
beats per minute | -4.40 (10.19) | -7.25 (14.43)

23. Primary Outcome: Average Change in Body Weight in Kilograms (kg) Comparing Baseline to Week 52.
Description: The subject's body weight was measured in kilograms(kg). The average value was calculated for each treatment group for the Baseline and Week 52 visits. The average change was determined by subtracting the average value at the Baseline Visit (Week 0) results from the Week 52 results (Week 52- Baseline (Week 0)).
  This measure was also collected as part of the study protocol at the Screening visit and Week 4, 8, 12, 16, 20, 24, 32 and 40.
Time Frame: At Baseline (Week0) and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 10 | 4
Kilograms | 4.59 (26.63) | 3.77 (9.49)

24. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Creatine Kinase (CK) Laboratory Values From Baseline to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant creatine kinase (CK) value if during the course of the study, they had at least one clinically significant CK result that was not present at baseline. Subjects had CK labs drawn at Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52.
Time Frame: At Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: Data for all subjects in the trial are not available for this assessment at all time points. One subject in the placebo group left the study before week 52. One subject in the etanercept group was lost to follow-up before the Week 52 visit.
  Data may also be missing due to the subject's refusal to complete an assessment or examiner error.
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 1 | 2

25. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Alanine Aminotransferase (ALT) Laboratory Values From Baseline to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not. A subject was considered to have a treatment emergent, clinically significant ALT value if during the course of the study, they had at least one clinically significant ALT result that was not present at baseline.
  Subjects had ALT labs drawn at Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52.
Time Frame: At Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 1 | 1

26. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Gamma-glutamyl Transpeptidase (GGT) Laboratory Values From Baseline to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant GGT value if during the course of the study, they had at least one clinically significant GGT result that was not present at baseline. Subjects had GGT labs drawn at Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52.
Time Frame: Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 0 | 1

27. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Aldolase Laboratory Values From Baseline to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant Aldolase value if during the course of the study, they had at least one clinically significant Aldolase result that was not present at baseline. Subjects had Aldolase labs drawn at Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52.
Time Frame: Screening, Baseline (Week0), Week 4, 8,12, 16, 20, 24, 32, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 1 | 2

28. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Glucose Laboratory Values From Baseline to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant Glucose value if during the course of the study, they had at least one clinically significant Glucose result that was not present at baseline. Subjects had Glucose labs drawn at Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52.
Time Frame: At Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 0 | 1

29. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Potassium Laboratory Values From Baseline to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant Potassium value if during the course of the study, they had at least one clinically significant Potassium result that was not present at baseline. Subjects had Potassium labs drawn at Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52.
Time Frame: Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 0 | 0

30. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal White Blood Cell Count (WBC) Values From Baseline to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant White Blood Cell (WBC) value if during the course of the study, they had at least one clinically significant WBC result that was not present at baseline. Subjects had WBC labs drawn at Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52.
Time Frame: Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 0 | 1

31. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Hemoglobin Laboratory Values From Baseline to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant Hemoglobin value if during the course of the study, they had at least one clinically significant Hemoglobin result that was not present at baseline. Subjects had hemoglobin labs drawn at Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52.
Time Frame: At Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 0 | 0

32. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Hematocrit Laboratory Values From Baseline to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant hematocrit value if during the course of the study, they had at least one clinically significant hematocrit result that was not present at baseline. Subjects had hematocrit labs drawn at Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52.
Time Frame: At Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 0 | 0

33. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Platelet Counts From Baseline to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant platelet value if during the course of the study, they had at least one clinically significant platelet result that was not present at baseline. Subjects had platelet labs drawn at Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52.
Time Frame: At Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 0 | 0

34. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Urine Leukocyte Values From Baseline to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant value if during the course of the study, they had at least 1 clinically significant urine leukocyte result that was not present at baseline. Subjects had urine leukocyte labs collected at Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52.
Time Frame: At Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 0 | 0

35. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Urine Protein Laboratory Values From Baseline to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant value if during the course of the study, they had at least one clinically significant urine protein result that was not present at baseline. Subjects had urine protein labs collected at Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52.
Time Frame: At Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 1 | 1

36. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Urine Glucose Laboratory Values From Baseline to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant value if during the course of the study, they had at least one clinically significant urine glucose result that was not present at baseline. Subjects had urine glucose labs collected at Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52.
Time Frame: At Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 0 | 1

37. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Urine Ketone Laboratory Values From Baseline to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant value if during the course of the study, they had at least one clinically significant urine ketone result that was not present at baseline. Subjects had urine ketone labs collected at Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52.
Time Frame: At Screening, Baseline (Week0), Week 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 0 | 0

38. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Serum 25-hydroxyvitamin D (25-OH VitD) Laboratory Values From the Screening Visit to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant value if during the course of the study, they had at least one clinically significant serum 25-hydroxyvitamin D (25-OH VitD) result that was not present at baseline. Subjects had 25-OH VitD labs collected at Screening and at the Week 52 visit.
Time Frame: Screening visit and Week 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 0 | 0

39. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Antinuclear Antibody Test (ANA) Values From the Screening Visit to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant value if during the course of the study, they had at least one clinically significant Antinuclear Antibody Test (ANA) result that was not present at baseline. Subjects had ANA labs collected at Screening, Week 12, 24, 40, and 52.
Time Frame: At Screening, Week 12, 24, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 1 | 0

40. Primary Outcome: Frequency of Subjects With Treatment Emergent, Clinically Significant, Abnormal Monoclonal Protein Detection by Serum Protein Electrophoresis (SPEP) From the Screening Visit to Week 52
Description: The site investigators used the reference ranges provided by the lab that completed the testing of the sample to determine if the value was abnormal. If a value was abnormal, the site investigator would determine if the value was clinically significant or not.
  A subject was considered to have a treatment emergent, clinically significant value if during the course of the study, they had at least one clinically significant monoclonal protein value that was not present at baseline. Subjects had monoclonal protein labs collected at Screening, Week 12, 24, 40, and 52.
Time Frame: Screening visit, Week 12, 24, 40, and 52
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
participants | 0 | 0

41. Primary Outcome: Average Cumulative Dosage of Prednisone Over the One Year Study Period
Description: The average cumulative dosage of prednisone over the one year period of the study was calculated. The results are presented by treatment group.
Time Frame: Baseline until week 52
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
mg | 5907.09 (3482.85) | 9917.65 (4762.09)

42. Secondary Outcome: Average Daily Dose of Prednisone From Baseline to Week 52
Description: The average daily dose of prednisone from baseline to week 52 was calculated by treatment group.
Time Frame: Baseline through Week 52
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 11 | 5
mg | 17.00 (9.92) | 36.40 (21.37)

ADVERSE EVENTS:
Time Frame: from screening to one month after completion of the study (at least 56 wks)
Arm/Group | Etanercept | Placebo
Serious Adverse Events (participants affected / at risk) | 3/11 | 3/5
Other Adverse Events (participants affected / at risk) | 11/11 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=11) | Placebo (N=5)
Partner Pregnant (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Post Herpetic Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Acute Psychosis (Psychiatric disorders) | 1 (2) | 0 (0)
Viral Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Dermatomyositis Flare (Nervous system disorders) | 0 (0) | 1 (1)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Etanercept (N=11) | Placebo (N=5)
Abdominal Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Distention (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anxiety/Mood Alternation (Psychiatric disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Auditory/Ear-Other- Tingling in ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Bladder Infection (Infections and infestations) | 0 (0) | 1 (1)
Bleeding- Vaginal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blurred Vision (Eye disorders) | 2 (2) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Burning sensation right foot (Nervous system disorders) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1)
Cataracts (Eye disorders) | 1 (2) | 0 (0)
Chest tightness (Cardiac disorders) | 0 (0) | 1 (1)
Chest tightness (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Cholesterol High (Investigations) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dental/Teeth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 3 (3)
Difficulty Swallowing (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1)
Dryness inner eyelids (Eye disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Edema: Left Knee Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Elevated Aldolase (Investigations) | 1 (1) | 1 (1)
Elevated ALT (Investigations) | 0 (0) | 1 (1)
Elevated AST (Investigations) | 0 (0) | 1 (1)
Elevated CK (Investigations) | 2 (2) | 1 (1)
Elevated GGT (Investigations) | 1 (1) | 1 (1)
Elevated Glucose (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Elevated WBC (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fall; Right Scalp Abrasion & Hematoma, R Chest Wall Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Fatty liver (Hepatobiliary disorders) | 0 (0) | 1 (1)
Fecal Urgency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 4 (5)
Heartburn (Gastrointestinal disorders) | 3 (4) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Increased Edema (Vascular disorders) | 0 (0) | 1 (1)
Increased Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Increased weakness right lower leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Infection- Sacral area (Infections and infestations) | 1 (1) | 0 (0)
Infection NOS (Viral Syndrome) (Infections and infestations) | 1 (1) | 0 (0)
Infection Upper Airway (Infections and infestations) | 5 (8) | 1 (1)
Infection with Normal ANC - Conjunctiva (Infections and infestations) | 1 (1) | 0 (0)
Infection with Normal - ANC - UTI (Infections and infestations) | 1 (1) | 0 (0)
Infection- Conjuctiva (Infections and infestations) | 1 (1) | 0 (0)
Infection - Lip (Infections and infestations) | 1 (1) | 1 (1)
Infection - Other (Gastrointestinal) (Infections and infestations) | 0 (0) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 0/0 (0) | 1 (1)
Injection Site Reaction (General disorders) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Interstital Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laboratory/Other- Abnormal PAP Smear (Investigations) | 1 (1) | 0 (0)
Left Antecubital Fossa Scab- Wound Complication - Noninfectious (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Left Kidney Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Low WBC Count (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Mechanics Hand on Right Index Finger- Hand/Foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Pains (Musculoskeletal and connective tissue disorders) | 6 (27) | 3 (4)
Nausea (Gastrointestinal disorders) | 3 (5) | 2 (4)
Neuropathy (Nervous system disorders) | 3 (3) | 1 (1)
Replacement of pacemaker (Surgical and medical procedures) | 0 (0) | 1 (1)
Ear numbness (Nervous system disorders) | 1 (1) | 0 (0)
Endometrial polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Increased Vit D Level (Investigations) | 0 (0) | 1 (1)
Pain- Ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pain- Throat/Pharynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Periungal Finger Infections (Infections and infestations) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin Burn Left Forearm Vent Surface (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin/Cellulitus Right Great Toe (Infections and infestations) | 1 (1) | 0 (0)
Spinal Headache (Nervous system disorders) | 1 (1) | 0 (0)
Stomach Cramps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subconjuctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Syndromes- Other (Sicca) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 3 (4) | 0 (0)
Transient Cardiac Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Urine Glucose Pos. (Investigations) | 0 (0) | 1 (1)
Urine Protein Pos. (Investigations) | 0 (0) | 1 (1)
UTI (Infections and infestations) | 1 (1) | 0 (0)
Viral Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Viral Hepatitis (Infections and infestations) | 1 (1) | 0 (0)
Vitamin D Low (Investigations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (3)
Worsening of Dermato (Nervous system disorders) | 1 (1) | 0 (0)
Worsening Skin Rash (Skin and subcutaneous tissue disorders) | 5 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No